CLINICAL TRIAL: NCT03118908
Title: Clinical Evaluation of Effectiveness and Safety of Combined Use of Dietary Supplements Amberen and Smart B by Women With Climacteric Syndrome
Brief Title: Clinical Evaluation of Effectiveness and Safety of Amberen and Smart B by Women With Climacteric Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Kuznetsova Irina, Chief Researcher, Scientific Research Centre, Women's Health Scientific Research Department, I.M. Sechenov First Moscow State Medical University, University hospital #2, Obstetrics and Gynecology clinic., I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AmberenSmartB-2017
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-07

CONDITIONS: Climacteric Syndrome; Menopause
Keywords: Succinate; B complex vitamins; menopause

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amberen and Smart B (Experimental): Amberen - a dietary supplement: 2 capsules (one while capsule 200 mg and one orange capsule 200 mg) are taken once a day with a meal, preferably after breakfast, for 3 months.
  SMART В - a dietary supplement: 1 capsule per day (166 mg) is taken once a day with a meal, preferably after breakfast, for 3 months, concurrently with Amberen.
  Interventions: Dietary Supplement: Amberen; Dietary Supplement: Smart B
- Placebo (Placebo Comparator): Placebo is taken as follows: 3 capsules (one while capsule 200 mg, one orange capsule 200 mg, one capsule 166mg) are taken once a day with a meal, preferably after breakfast, for 3 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Amberen — Amberen is a succinate-based dietary supplement previously shown to help provide relief for common menopausal symptoms.
  Arms: Amberen and Smart B
Dietary Supplement: Smart B — Smart B contains vitamins B1, B2, B6, B9, B12 and sodium fumarate.
  Arms: Amberen and Smart B
Dietary Supplement: Placebo — Placebo capsules are identical to Amberen and Smart B capsules.
  Arms: Placebo

SUMMARY:
To evaluate effectiveness and safety of combined use of dietary supplements Amberen and Smart B by women with a typical (without complications) form of climacteric syndrome, with mild to moderate symptoms.

DETAILED DESCRIPTION:
1. To evaluate effectiveness of combined use of dietary supplements Amberen and Smart B (vs placebo) by women with a typical (without complications) form of climacteric syndrome, with mild to moderate vegetative symptoms during perimenopause and menopause in regards to vasomotor, endocrine-metabolic, and neuro-psychological dysfunctions;
2. To evaluate safety of combined use of dietary supplements Amberen and Smart B (vs placebo) by women with a typical (without complications) form of climacteric syndrome, with mild to moderate vegetative symptoms during perimenopause and menopause, lasting no less than 1 year in regards to vasomotor, endocrine-metabolic, and neuro-psychological dysfunctions;
3. To develop recommendations for combined use of dietary supplements Amberen and Smart B for women with a typical (without complications) form of climacteric syndrome, with mild to moderate vegetative symptoms during perimenopause and menopause (menopausal for at least 1 year).

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 42-60 years of age;
* Patient with diagnosis of "climacteric syndrome", in typical or non-complicated form, mild or moderate vegetative symptoms during menopause i.e. absence of menstrual period for at least 1 year;
* Ability to read and understand informed consent form for the study's participation;
* Patients without risk factors and changes in the breast tissue based on the mammogram;
* Patients with medical history of risk factors without changes in the breast tissue;
* Ability to adhere to the conditions of the study.

Exclusion Criteria:

* Presence of female reproductive system cancers (breast cancer, cervical cancer etc.);
* Presence of extragenital oncological conditions, except those in complete remission for 5 years or more;
* Conditions requiring emergency or planned hospitalization in the next 6 months;
* Presence of hormonally-active extragenital endocrine diseases (thyroid, adrenal, pituitary, hypothalamus);
* Surgical interventions done on sex organs or breasts, 1 year or less prior to the screening;
* Any surgeries done less than 3 months prior to the screening;
* Patients receiving HRT;
* Psychiatric conditions;
* Diabetes;
* Total ovariectomy
* Patients taking any other dietary supplements that can affect climacteric syndrome within the last month before enrolling in the study

  * High risk of non-compliance

Ages: 42 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 107 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Spilberger-Hanin (Situational anxiety) | week 12
  The decrease of situational anxiety, measured as statistically significant reduction of the score in corresponding subscale
Spilberger-Hanin (Personal anxiety) | week 12
  The decrease of personal anxiety, measured as statistically significant reduction of the score in corresponding subscale
Spilberger-Hanin (Actual anxiety) | week 12
  The decrease of actual anxiety, measured as statistically significant reduction of the score in corresponding subscale. Actual anxiety as a sum of situational and personal anxiety scores was introduced by Hanin in his modification of original State-Trait Anxiety Inventory.
WELL-BEING, LEVEL OF ACTIVITY, MOOD QUESTIONNAIRE (well-being) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
WELL-BEING, LEVEL OF ACTIVITY, MOOD QUESTIONNAIRE (activity) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
WELL-BEING, LEVEL OF ACTIVITY, MOOD QUESTIONNAIRE (mood) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
Anxiety (measured by Hospital Anxiety and Depression Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
Depression (measured by Hospital Anxiety and Depression Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms

SECONDARY OUTCOMES:
"Heart beating quickly and strongly" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling tense or nervous" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Difficulty in sleeping" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Excitable" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Attacks of panic" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Difficulty in concentrating" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling tired or lacking in energy" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Loss of interest in most things" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling unhappy or depressed" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Crying spells" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Irritability" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Feeling dizzy or faint" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Pressure or tightness in head or body" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Parts of body feeling numb or tingling" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Headaches" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Muscle or joint pains" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Loss of feeling in hands or feet" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
Breathing difficulties" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Hot flushes" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Sweating at night" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
"Loss of interest in sex" symptom (Greene Climacteric Scale) | week 12
  Statistically significant reduction in designated symptom severity, compared between arms
Blood plasma estradiol levels, pg/ml | week 12
  Statistically significant reduction in the levels, compared between arms
Weight, kg | week 12
  Statistically significant reduction in the measurement, compared between arms

CONTACTS AND LOCATIONS:
Locations (1):
- Sechenov First Moscow Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No